CLINICAL TRIAL: NCT00736723
Title: NT-proBNP in Postoperative/Posttraumatic Critically Ill Patients With Severe SIRS/Sepsis and Shock
Brief Title: NT-proBNP in ICU Postoperative/Posttraumatic Patients With Shock
Acronym: NICUPS
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, MBA, University of Ulm
Other Study IDs: Anae_ICU_Ulm_NT-proBNP
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: SIRS; Sepsis; Shock; Critically Ill; Multiple Organ Dysfunction Syndrome
Keywords: NT-proBNP; myocardial dysfunction; humans; patients; polytrauma; complement; inflammation; inflammatory response; biomarkers; cytokines; cell surface markers; functional polymorphisms; infections; systemic inflammatory response syndrome; SIRS; sepsis; severe sepsis; shock; organ dysfunctions; SOFA; severity of disease; APACHEII; SAPSII; SPAPS3; length of stay; outcome; mortality
MeSH Terms: conditions — Sepsis; Shock; Critical Illness; Multiple Organ Failure; Multiple Trauma; Inflammation; Infections; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients non-septic shock: Postoperative/posttraumatic critically ill patients with non-septic shock
- Patients septic shock: Postoperative/posttraumatic critically ill patients with septic shock

SUMMARY:
The purpose of this study is to determine the course of NT-proBNP plasma concentrations in the context of confounding parameters in postoperative/posttraumatic critically ill patients with severe SIRS/sepsis and shock.

DETAILED DESCRIPTION:
In the recent sepsis-definitions, myocardial depression is included in the definition of severe sepsis, indicated as lowered cardiac index or echocardiographically documented cardiac dysfunction. Myocardial dysfunction occurs in greater than 50% of patients with severe sepsis and septic shock. In this context, B-type natriuretic peptid (BNP) from ventricular myocytes may serve as a surrogate biomarker for the evaluation and quantification of myocardial dysfunction. Biologically active BNP is cleaved into inactive NT-proBNP, which is supposed to be a better marker of myocardial dysfunction and prognosis in patients with severe sepsis and septic shock. However, severity of illness dependent association of myocardial dysfunction, especially left ventricular diastolic function, dosage of norepinephrine, NT-proBNP and biomarker plasma concentrations has not been systematically investigated in postoperative/posttraumatic patients in septic shock or volume-deficiency/hemorrhagic shock. Moreover, data regarding NT-proBNP plasma concentrations and renal function in postoperative/posttraumatic patients are sparse. Therefore, this prospective observational study will enroll n= 200 postoperative/posttraumatic patients to monitor longitudinally NT-proBNP, biomarkers, and cell surface markers on leukocytes to find out whether there is a discriminating pattern of myocardial dysfunction, NT-proBNP and biomarkers in patients with non-septic or septic shock, respectively, and with beneficial or harmful outcome.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill, postoperative/posttraumatic patients with severe systemic inflammatory response syndrome (SIRS) or severe sepsis

Exclusion Criteria:

* Life expectancy < 24 hours
* Participation in other trials
* Known or suspected pregnancy
* Contraindications for transesophageal echocardiography (TEE): severe disease of the esophagus (hernia, strictures, esophageal resection, severe bleeding disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative/posttraumatic critically ill patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, MBA, Principal Investigator — Clinic of Anesthesiology, University Hospital Medical School, Steinhoevelstrasse 9, 89070 Ulm, Germany
Locations (1):
- Clinic of Anesthesiology, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss M, Huber M, Nass M, Huber-Lang M, Koenig W, Schneider M. NT-proBNP and HMGB1 in surgical critically ill patients with hypovolemic or septic shock.Infection Suppl. II September 2011; 39: S116-117 5th International Congress of the German Sepsis Society, Weimar Sepsis Update Bridging The Gap, Weimar, 07. - 10.09.2011.
- [Result] Weiss M, Huber M, Nass M, Huber-Lang M, Koenig W, Schneider M. NT-proBNP serum concentrations in surgical critically ill patients with non-septic and septic shock. INNOVATIVE JOURNAL OF MEDICAL AND HEALTH SCIENCE 3 (4): 177-184, 2013.

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Non-septic Shock: critically ill surgical patients admitted from 01 July 2008 to 31 Dec 2008 in the ICU revealing non-septic shock
- Patients With Septic Shock: critically ill surgical patients admitted from 01 July 2008 to 31 Dec 2008 in the ICU revealing septic shock
Period: Overall Study
Arm/Group | Patients With Non-septic Shock | Patients With Septic Shock
Started | 30 | 21
Completed | 26 | 18
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: surveyed daily for sepsis, organ dysfunctions and shock
Groups:
- Postoperative/Posttraumatic Patients With Non-septic Shock: Postoperative/posttraumatic critically ill patients with non-septic shock
- Postoperative/Posttraumatic Patients With Septic Shock: Postoperative/posttraumatic critically ill patients with septic shock
- Total: Total of all reporting groups
Arm/Group | Postoperative/Posttraumatic Patients With Non-septic Shock | Postoperative/Posttraumatic Patients With Septic Shock | Total
Number analyzed (Participants) | 26 | 18 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 10 | 8 | 18
Age, Continuous [Median (Full Range); unit: years] | 53 [20 to 80] | 60 [37 to 88] | 57 [20 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  Germany | 26 | 18 | 44

OUTCOME MEASURES:

1. Primary Outcome: Pattern of NT-proBNP, Biomarkers and Surface Markers on Leukocytes
Description: maximal NT-proBNP concentrations in critically ill surgical patients admitted from 01 July 2008 to 31 Dec 2008 in the ICU revealingnonseptic and septic shock
Time Frame: 01 July 2008 to 31 Dec 2008
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Patients Non-septic Shock | Patients Septic Shock
Number analyzed (Participants) | 26 | 18
pg/ml | 902 [39 to 31,937] | 4,429 [193 to 35,000]

ADVERSE EVENTS:
Groups:
- Hypovolemic Shock: Shock was defined as hypotension despite adequate volume resuscitation without infection, a systolic blood pressure of < 90 mmHg, or the need of vasopressors to keep blood pressure ≥ 90 mmHg. 26 patients.
- Septic Shock: Shock was defined as hypotension despite adequate volume resuscitation due to infection, a systolic blood pressure of < 90 mmHg, or the need of vasopressors to keep blood pressure ≥ 90 mmHg. 18 patients.
Arm/Group | Hypovolemic Shock | Septic Shock
All-Cause Mortality (participants affected / at risk) | 2/26 | 3/18
Serious Adverse Events (participants affected / at risk) | 2/26 | 3/18
Other Adverse Events (participants affected / at risk) | 0/26 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypovolemic Shock (N=26) | Septic Shock (N=18)
Death (Immune system disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Myocardial depression has not been verified in our patients by a low cardiac index or by echocardiography

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No